CLINICAL TRIAL: NCT04985071
Title: Study of Pancreatic Fistula and Bleeding Complication After Pancreaticoduodenectomy in Treatment Periampullary Cancer
Brief Title: Complication of Pancreatic Fistula and Bleeding After Pancreaticoduodenectomy in Treatment Periampullary Cancer
Acronym: PF
Status: Completed | Type: Observational
Sponsor: Vo Truong Quoc (Other)
Responsible Party: Sponsor-Investigator, Vo Truong Quoc, General Surgery Department, Principal Investigator, Clinical Professor, University of Medicine and Pharmacy at Ho Chi Minh City
Organization: University of Medicine and Pharmacy at Ho Chi Minh City (Other)
Other Study IDs: VTrQuoc
Record Dates: First submitted 2021-07-26; First posted 2021-08-02 (Actual); Last update posted 2024-05-13 (Actual); Status verified 2024-05

CONDITIONS: Periampullary Cancer; Pancreatic Fistula; Bleeding
Keywords: Pancreatic Surgery
MeSH Terms: conditions — Pancreatic Fistula; Hemorrhage | interventions — Pancreaticoduodenectomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 90 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Pancreaticoduodenectomy — Patient with periampullary cancer will be underwent pancreaticoduodenectomy in 2 types of pancreatic-jejunal anastomosis reconstructions. We describe the postoperative complications (pancreatic fistula and bleeding) and analysis the risk factors relate to those complications
  Other Names: Medical treatment after operation

SUMMARY:
This multi-site study will be done across Hepatobiliary and Pancreatic Surgery Department at Cho Ray Hospital and University and Pharmacy Center. Patients who are diagnosed with periampullary cancer from August 2021 to August 2023 will be underwent pancreaticoduodenectomy. We will follow-up for their pancreatic fistula and bleeding complication and analysis some risk factors.

DETAILED DESCRIPTION:
The investigator will conduct this study at both site at the same time: Cho Ray Hospital and University and Pharmacy Center. The investigator will directly consult the patient to participate in the study, collect the preoperative information, intraoperative protocol and postoperative data. The investigator will statically analysis the incident of the morbidity (mainly for pancreatic fistula and bleeding), and invest some risk factors relating to those complications.

Plan for conducting the study:

* The patient diagnosed with periampullary cancer will be consulted with surgical method, operative risks, postoperative complications and agree to participate in the study. The patient signes a consent form to participate in the study.
* Pancreaticoduodenectomy will be performed according to the uniformity protocol of both hospitals: Cho Ray Hospital and University of Medicine and Pharmacy Center.
* Post-operative data will be collected and based on the general procedure.

Data analysis

* To determine the incidence of pancreatic fistula and bleeding, survival analysis will be used.
* To determine the association of risk factors with pancreatic fistula and bleeding, logistic regression was used, the value with p < 0.05 will be included in the multivariable regression model to determine the real risk factors.

Sample size:

• The investigator expect approximately 100 patients in the first year in both centers. And the investigator hope at least 110 patients in the whole conducting time.

Plan for missing data:

• The investigator will directly collect the patient information before the operation, observe the operation process and follow-up the postoperative during. Investigator will remove any case that missing preoperative information, operative data or post-operative laboratory test.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with periampullary cancer meet the following criteria:

  * Possibility to perform pancreaticoduodenectomy based on preoperative imaging and intraoperative exploration.
  * The postoperative pathology is adenocarcinoma (of the ampulla of Vater, common bile duct, duodenum or pancreas)

Exclusion Criteria:

* The patient has other organ's cancer beyond periampullary cancer.
* Patient's medical conditions contraindicate for anesthesia.
* The patient does not consent to participate in the study

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with periampullary cancer will be underwent pancreaticoduodenectomy and will be followed-up after operation.
Sampling Method: Probability Sample
Enrollment: 183 (Actual)
Dates: Start 2021-08-01 (Actual); Primary Completion 2023-10-31 (Actual); Study Completion 2023-10-31 (Actual)

PRIMARY OUTCOMES:
Pancreatic fistula | 90 post-operative days
  Rate of post-operative pancreatic fistula, risk factors associate to pancreatic fistula

SECONDARY OUTCOMES:
Bleeding complication | 90 post-operative days
  Rate and location of post-operative bleeding, risk factors relate to this complication

CONTACTS AND LOCATIONS:
Overall Officials: TruongQuoc Vo, Doctor, Principal Investigator — University of Medicine and Pharmacy at HoChiMinh City
Locations (1):
- Phan Minh Tri, Ho Chi Minh City, Vietnam

IPD SHARING:
Plan to Share IPD: No
The IPD will be saved as a excel and spss file (with a password to open). This data can be shared with other researchers if needed.

REFERENCES:
- [Result] Melloul E, Lassen K, Roulin D, Grass F, Perinel J, Adham M, Wellge EB, Kunzler F, Besselink MG, Asbun H, Scott MJ, Dejong CHC, Vrochides D, Aloia T, Izbicki JR, Demartines N. Guidelines for Perioperative Care for Pancreatoduodenectomy: Enhanced Recovery After Surgery (ERAS) Recommendations 2019. World J Surg. 2020 Jul;44(7):2056-2084. doi: 10.1007/s00268-020-05462-w. PMID 32161987
- See also: Guidelines for Perioperative Care for Pancreaticoduodenectomy — https://pubmed.ncbi.nlm.nih.gov/32161987/